CLINICAL TRIAL: NCT07044206
Title: Prospective Randomized Comparative Study of Interbody Bone Fusion Between Two Osteoinductive Bioactive Bone Substitutes After Anterior Lumbar Interbody Arthrodesis in Degenerative Lumbar Disc Surgery in Adults
Brief Title: Comparaison of Interbody Bone Fusion Between Two Osteoinductive Bioactive Bone Substitutes After Anterior Lumbar Interbody Arthrodesis in Degenerative Lumbar Disc Surgery in Adults
Acronym: FUSALIF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECHMPL23_0450
Record Dates: First submitted 2025-06-16; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Disc Degeneration
Keywords: spinal surgery; spinal fusion; intervertebral disc
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group : Interbody fusion with bone substitute Magnetos Putty, Kuros medical (Experimental): Subjects randomly assigned to the intervention group will benefit from Magnetos Putty, Kuros during surgery
  Interventions: Device: Use of bone substitute during intervertebral fusion surgery
- Control group : Interbody fusion with conventional bone substitute GlassBone Putty, Noraker (Active Comparator): Subjects randomly assigned to the control group will benefit from GlassBone Putty, Noraker during surgery
  Interventions: Device: Use of bone substitute during intervertebral fusion surgery

INTERVENTIONS:
Device: Use of bone substitute during intervertebral fusion surgery — Participants randomized will receive bone substitute during intervertebral fusion surgery. Routine postoperative follow-up procedure (identical for both groups) with two postoperative visits at 3 months and 12 months.

SUMMARY:
Disc degeneration is a progressive deterioration process of the intervertebral disc, which can manifest as significant low back pain and a loss of mobility that interferes with daily activities. This condition is naturally age-related and exacerbated by traumatic events, lifestyle factors, and individual genetic susceptibilities. Treatment for advanced disc degeneration typically involves surgery (spinal fusion) aimed at addressing and fusing the affected intervertebral discs using an interbody implant combined with a bone graft.

Although the use of interbody implants promotes temporary fusion, long-term success largely depends on the bone substitute used, with failure rates ranging from 10 to 20% (unsuccessful fusion, persistent symptoms, need for reoperation). Historically, autologous bone grafting was the standard, but it carries disadvantages related to pain and invasiveness. Synthetic, bioactive bone substitutes are now used, although their effectiveness varies.

Animal studies support the hypothesis that a new substitute based on specific osteo-immunology technology (MagnetOs, Kuros) could offer superior results compared to autologous bone grafts and competing osteo-inductive materials, while being minimally invasive. This study aims to evaluate its properties in terms of bone fusion and its impact on functional scores in patients, hypothesizing a significant improvement in fusion rates and functional scores with this new substitute.

DETAILED DESCRIPTION:
Degenerative lumbar spine disease increasingly relies on surgery to treat and fuse one or more pathological intervertebral discs. The transabdominal retroperitoneal, or anterior, approach allows full access to and treatment of the diseased disc, enabling a more physiological restoration of spinal alignment. Implants placed in the interbody position provide immediate vertebral stabilization, while the bone graft or bone substitute added to the interbody implant enables long-term fusion through neo-ossification of the segment.

The quality and speed of fusion achieved largely depend on the bone substitute used, and this fusion is a key factor in obtaining good functional outcomes for the patient. In approximately 10 to 20% of cases, this fusion does not succeed, resulting in persistent pain symptoms and potentially requiring reoperation.

Historically, to achieve this fusion, autologous bone was harvested from another anatomical site, most often the iliac crest. This autologous bone graft requires an additional incision, which is often associated with pain and discomfort. For these reasons, synthetic or biologic bone substitutes have been developed by pharmaceutical engineering to avoid bone harvesting, and are now routinely used in clinical practice.

To date, many bioactive bone substitutes have obtained marketing authorization, but their effectiveness varies depending on their physicochemical composition. It is accepted that the fusion rate could improve by up to 60% depending on the bone substitute used.

Animal studies support the hypothesis that a new bone substitute, referred to here as Substitute A, based on specific osteoimmunology technology (MagnetOs, Kuros), is equivalent to the current gold standard (autologous bone graft) in terms of achieved fusion, and superior to competing osteoinductive products that are routinely used at Montpellier University Hospital and in most other hospitals to achieve spinal fusion (6). This suggests the possibility of achieving equivalent outcomes through a faster, less invasive, less painful procedure with no limitation on the volume of substitute used.

Due to its favorable characteristics, this product (Substitute A) was recently endorsed by the Commission for Medicines and Sterile Medical Devices (CMDMS) of Montpellier University Hospital, authorizing its appropriate use in this indication, though currently limited to a small number of batches. This project would allow us to demonstrate the benefits of Substitute A so that it could subsequently be adopted for routine use.

This trial is a single-center, prospective, randomized, controlled superiority trial, with single-blind evaluation of the primary outcome measure. This study aims to include 100 patients. A non-stratified randomization with random block sizes will be performed to allocate participants in a 1:1 ratio into the following groups: Group A receiving the investigational device (bone substitute, Magnetos Putty, Kuros Medical) and Group B receiving the routine treatment (bone substitute, GlassBone Putty, Noraker).

Simplified study calender:

Visit 1: Information between 6 months and 1 month before Day 0 Preoperative consultation to determine the indication for surgery and the date of the operation

* Presentation of the trial, description of the practical aspects of the study and randomization process
* Provision of the information sheet

Visit 1: Before the intervention (Day -1) Re-presentation of the trial, description of the practical aspects of the study and randomization process

* Verification of eligibility criteria
* Obtaining informed consent
* Collection of demographic data : age, sex, occupation, Body Mass Index (BMI), medication use, smoking, alcohol consumption, medical history)
* Health questionnaires : Visual Analogue Scale (VAS), Oswestry Disability Index (ODI)
* Collection of imaging data : high-resolution lumbar Computed Tomography (CT) scan and lumbar X-ray)

Visit 2: Day 0 (Surgical intervention day) Randomization will be performed at the earliest, the day before or on the day of the intervention.

Patients will be randomized into either the conventional or experimental arm. The allocated arm will be communicated to the neurosurgeon investigator responsible for the operation. The patient will remain blinded to their treatment group.

The surgical intervention will be performed according to the standard anterior lumbar fusion procedure, except for the bone substitute, which will vary according to randomization.

Visit 3: 3 months (+/- 15 days)

Following the usual care for patients who have undergone anterior lumbar interbody fusion:

* Low back and radicular pain (VAS)
* Functional score (ODI)
* Imaging for a 3-month assessment (high-resolution lumbar CT scan)
* Collection of additional data (return to work, medication use)

Visit 4: 12 months (+/- 15 days)

Following the usual care for patients who have undergone anterior lumbar interbody fusion:

* Low back and radicular pain (VAS)
* Functional score (ODI)
* High-resolution lumbar CT scan and lumbar X-ray in weight-bearing and dynamic positions
* Collection of additional data (return to work, medication use...)

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years inclusive
* Oswestry Disability Index (ODI) >25
* Chronic low back pain and/or radicular pain lasting for more than 6 months
* Failure of medical and rehabilitative treatment
* Patient presenting with one of the following: grade 1 degenerative spondylolisthesis without isthmic lysis, or disc degeneration, or mixed pathology (degeneration and lumbar stenosis)
* Patient eligible for anterior approach spinal fusion surgery with interbody cage

Exclusion Criteria:

* History of spinal surgery at the lumbar level, excluding isolated discectomies for disc herniation
* Confirmed osteoporosis
* Surgical fusion at an adjacent level
* Contraindication to Magnetos Putty or GlassBone Putty:

  1. Use of medications interfering with calcium metabolism
  2. Severe systemic or metabolic bone disorders affecting bone healing or lesions
  3. Untreated acute or chronic infection requiring appropriate therapy
  4. Patients with severe trauma and open external wounds near the defect site, at risk of infection
  5. Known allergy to bioactive glass or its components (Ca2+, PO43-, Na+, and Si(OH)4), polyethylene glycol, and/or glycerol
  6. Patients who have undergone or will undergo chemotherapy or radiotherapy at or near the implantation site
  7. Severe renal or hepatic infections
  8. Unrepaired dural tear in craniospinal surgery
* Patients requiring placement of more than one implant
* Subject unable to read and/or write fluent French, or illiterate
* Subject already participating in another interventional clinical trial that could interfere with this study
* Uncontrolled psychiatric illness
* Lack of written informed consent after a reflection period
* Individuals with a dependency or employment relationship with the sponsor or investigator
* Subject enrolled in another study with an ongoing exclusion period (Article L1121-12)
* Subject not affiliated with or not a beneficiary of the French social security system (L1121-8-1)
* Protected populations under French Public Health Code:

  1. Pregnant or breastfeeding women (L. 1121-5)
  2. Individuals deprived of liberty (art. L. 1121-6) (by judicial, administrative decision or involuntary hospitalization)
  3. Protected adults (under guardianship, curatorship, or legal protection) (L. 1121-8)
* Women planning to become pregnant within the year

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in the Oswestry Disability Index (ODI) score from baseline (preoperative assessment) to 12 months following lumbar spinal fusion surgery for disc degeneration in adult patients. | Baseline to 12 months post-surgery
  The primary efficacy endpoint will assess functional disability improvement by measuring the variation in ODI score between the preoperative evaluation and the 12-month postoperative follow-up. The ODI is a self-administered questionnaire used to assess the degree of disability related to low back pain. It consists of 10 sections, each scored from 0 to 5, resulting in a total score ranging from 0 (no disability) to 50 (maximum disability).

SECONDARY OUTCOMES:
Assessment of interbody fusion at 12 months using CT scan. | 12 months post-surgery
  The assessment of fusion grade is performed in a blinded manner by two trained readers (a neuroradiologist and a neurosurgeon), based on consensus. Evaluation is conducted using a high-resolution (millimetric) lumbar CT scan performed 12 months after the surgical procedure.
  The results are classified into three grades: definite fusion, uncertain fusion, and definite pseudarthrosis.
Evaluation of pain and functional disability using Visual Analog Scale (VAS) for low back and radicular pain at 3 and 12 months postoperatively. | 3 months and 12 months post-surgery
  Pain intensity will be assessed using the Visual Analog Scale (VAS) for both low back and radicular pain. This score will be recorded at 3-month and 12-month follow-up visits to evaluate the evolution of symptoms over time. The VAS is a patient-reported measure used to quantify pain intensity ranging from 0 to 10. A score of 0 indicates no pain, a score of 10 represents the worst possible pain.
Oswestry Disability Index (ODI) at 3 and 12 months. | 3 months and 12 months post-surgery
  Functional disability will be measured using the Oswestry Disability Index (ODI). This score will be recorded at 3-month and 12-month follow-up visits to evaluate functional recovery over time.
Use of analgesic and anti-inflammatory medications (steroidal and non-steroidal) at 3 and 12 months postoperatively. | 3 months and 12 months post-surgery
  Evaluation of postoperative consumption of pain medications, including steroidal and non-steroidal anti-inflammatory drugs (NSAIDs), at the 3-month and 12-month follow-up visits.
Rate of patient return to work at 3 and 12 months postoperatively | 3 months and 12 months post-surgery
  Rate of patient return to work at 3 and 12 months postoperatively. In cases where the patient has not returned to work, the reason for non-return will be documented.
Time to resumption of activity within 12 months | From surgery to 12 months postoperatively
  Time to resumption of activity within 12 months
Rate of re-hospitalization within 3 months following the surgical intervention. | Within 3 months post-surgery
  Rate of any unplanned hospital readmissions occurring within 3 months after the initial lumbar fusion surgery. The reason for each re-hospitalization will be recorded.
Reoperation at the initial surgical site during the 12-month follow-up period. | Within 12 months post-surgery
  Assessment of any surgical reintervention performed at the same anatomical site as the initial lumbar fusion within the 12-month follow-up period. The indication for reoperation will be documented (e.g., pseudarthrosis, infection, hardware failure...).

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Montpellier, Montpellier, France, France

IPD SHARING:
Plan to Share IPD: Undecided